CLINICAL TRIAL: NCT05903222
Title: The Effect of Posterior Pericardiotomy on the Incidence of Atrial Fibrillation After Cardiac Surgery - Extended Follow-Up (PALACS-EF) Study
Brief Title: The Effect of Posterior Pericardiotomy on the Incidence of Atrial Fibrillation After Cardiac Surgery-Extended Follow-Up
Acronym: PALACS-EF
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1502015867-Extension
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: postoperative; left posterior pericardiotomy; prevention; cardiac surgery
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Posterior Pericardiotomy: All patients who were randomized to receive posterior pericardiotomy (intervention) in the original PALACS trial.
  Interventions: Other: Non-Interventional
- No Posterior Pericardiotomy (control): All patients who were randomized to receive no intervention/no posterior pericardiotomy in the original PALACS trial

INTERVENTIONS:
Other: Non-Interventional — This study is a non-interventional study of all patients previously enrolled in the PALACS trial
  Groups: Posterior Pericardiotomy

SUMMARY:
The purpose of the Effect of Posterior Pericardiotomy on the Incidence of Atrial Fibrillation After Cardiac Surgery (PALACS, NCT02875405) trial was to determine if performing posterior left pericardiotomy at the time of cardiac surgery prevents atrial fibrillation after cardiac surgery. The purpose of the Posterior left pericardiotomy for the prevention of AtriaL fibrillation After Cardiac Surgery-Extended Follow-Up (PALACS-EF) study is to evaluate the effect of posterior left pericardiotomy on 5-year clinical outcomes.

DETAILED DESCRIPTION:
Post-operative atrial fibrillation (POAF) is a common complication of cardiac surgery which is observed in 30-40% of patients. POAF has also been associated with stroke, systemic embolism or cardiac failure during the years after surgery. Several strategies aimed at reducing the incidence of POAF have been investigated, including beta-blockers, amiodarone, and statins, with unsatisfactory results. In the randomized prospective clinical trial, the PALACS trial, 420 patients were randomized either to the intervention group, which received left posterior pericardiotomy at time of cardiac surgery, or to the control group, which did not receive posterior left pericardiotomy at time of cardiac surgery. Posterior left pericardiotomy was associated with a reduction in the incidence of POAF after surgery, but not with improvement in 30-day patient outcomes.

This non-interventional, prospective study is an extension follow-up study (PALACS-EF) of all patients who were enrolled in the original PALACS trial. It is designed to evaluate differences in clinical outcomes between patients who received posterior left pericardiotomy (intervention) versus those who did not (control) at median follow-up of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* This study will include all the subjects enrolled in the PALACS trial

Exclusion Criteria:

* Not enrolled in the PALACS trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in the PALACS trial
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-10-13 (Actual)

PRIMARY OUTCOMES:
Time to first occurrence of the composite of all-cause mortality and hospital readmission for cardiovascular causes | Median five-year follow-up

SECONDARY OUTCOMES:
Time to first occurrence of the composite of all-cause mortality and all-cause hospital readmission | Median five-year follow-up
Number of Adverse Events | Median five-year follow-up
  The following adverse events will be included in the count: Myocardial infarction, stroke, transient ischemic attack, new arrhythmia (atrial fibrillation versus non-atrial fibrillation), heart failure, systemic embolism

CONTACTS AND LOCATIONS:
Overall Officials: Leonard N Girardi, MD, Principal Investigator — Weill Cornell Medical College New York Presbyterian Hospital; Mario Gaudino, MD, Study Chair — Weill Cornell Medical College New York Presbyterian Hospital
Locations (1):
- Weill Cornell Medical College Department of Cardiothoracic Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biancari F, Mahar MA. Meta-analysis of randomized trials on the efficacy of posterior pericardiotomy in preventing atrial fibrillation after coronary artery bypass surgery. J Thorac Cardiovasc Surg. 2010 May;139(5):1158-61. doi: 10.1016/j.jtcvs.2009.07.012. Epub 2009 Aug 18. PMID 19691996
- [Background] Kaleda VI, McCormack DJ, Shipolini AR. Does posterior pericardiotomy reduce the incidence of atrial fibrillation after coronary artery bypass grafting surgery? Interact Cardiovasc Thorac Surg. 2012 Apr;14(4):384-9. doi: 10.1093/icvts/ivr099. Epub 2012 Jan 9. PMID 22235005
- [Background] Gaudino M, Sanna T, Ballman KV, Robinson NB, Hameed I, Audisio K, Rahouma M, Di Franco A, Soletti GJ, Lau C, Rong LQ, Massetti M, Gillinov M, Ad N, Voisine P, DiMaio JM, Chikwe J, Fremes SE, Crea F, Puskas JD, Girardi L; PALACS Investigators. Posterior left pericardiotomy for the prevention of atrial fibrillation after cardiac surgery: an adaptive, single-centre, single-blind, randomised, controlled trial. Lancet. 2021 Dec 4;398(10316):2075-2083. doi: 10.1016/S0140-6736(21)02490-9. Epub 2021 Nov 14. PMID 34788640
- [Derived] Gaudino M, Harik L, Redfors B, Sandner S, Alexander JH, Di Franco A, Dimagli A, Weinsaft J, Perezgrovas-Olaria R, Soletti GJ, Lau C, Mack C, Girardi L. The Effect of Posterior Pericardiotomy on the Incidence of Atrial Fibrillation After Cardiac Surgery-Extended Follow-Up study (PALACS-EF): rationale and design. Eur Heart J Open. 2023 Nov 17;3(6):oead118. doi: 10.1093/ehjopen/oead118. eCollection 2023 Nov. PMID 38035038
- See also: Weill Cornell Department of Cardiothoracic Surgery — https://ctsurgery.weillcornell.org/